CLINICAL TRIAL: NCT06628947
Title: A Phase II, Randomised, Controlled, Double Masked, Multiple Dose Study of the Safety, Tolerability and Efficacy of Intravitreal KIO-301 in Patients With Late-stage Retinitis Pigmentosa
Brief Title: A Phase II Study of Intravitreal KIO-301 in Patients With Late-stage Retinitis Pigmentosa
Acronym: ABACUS-2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kiora Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KIO-301-2101
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-07

CONDITIONS: Retinitis Pigmentosa
Keywords: Late-stage RP with No Light Perception; Late-stage RP with Low Vision
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Cohort design:
  Cohort 1A:
  • RP who have NLP will be randomised (2:1) to receive 50 μg KIO-301 or placebo
  Cohort 1B:
  • RP who have LV will be randomised (2:1) to receive 50 μg KIO-301 or placebo
  Cohort 2A:
  • RP who have NLP will be randomised (2:1) to receive 100 μg KIO-301 or placebo
  Cohort 2B:
  • RP who have LV will be randomised (2:1) to receive 100 μg KIO-301 or placebo
  Cohort 3A:
  • RP who have NLP will be randomised (2:1) to receive 25 μg KIO-301 or placebo
  Cohort 3B:
  • RP who have LV will be randomised (2:1) to receive 25 μg KIO-301 or placebo
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: This is a double masked study. As there is a colour difference between KIO-301 and placebo, (investigational medicinal product (IMP) administration will be performed by an unmasked dose administrator. The dose administrator will not discuss treatment administered with any other study staff, participants, or sponsor representatives, and will not conduct any other study activities or participant assessments.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 50 μg KIO-301 (Experimental): 50 μg KIO-301 or placebo administered by IVT injection bilaterally (OU) once every 6 weeks for 3 administrations per participant.
  Interventions: Other: Placebo (Sterile Saline or Balanced Salt Solution); Drug: 50 μg KIO-301
- 100 μg KIO-301 (Experimental): 100 μg KIO-301 or placebo administered by IVT injection OU once every 6 weeks for 3 administrations per participant.
  Interventions: Other: Placebo (Sterile Saline or Balanced Salt Solution); Drug: 100 μg KIO-301

INTERVENTIONS:
Other: Placebo (Sterile Saline or Balanced Salt Solution) — A control 50 μl injection of clear sterile saline or balanced salt solution (BSS) liquid.
Drug: 100 μg KIO-301 — KIO-301 drug product is an ophthalmic formulation of the drug substance KIO-300-Cl in sulfobutylether-β-cyclodextrin, sucrose, phosphate buffer salts and water suitable for IVT injection. The drug substance KIO-300-Cl is a quaternary ammonium chloride salt of the active compound KIO-300.
  Arms: 100 μg KIO-301
Drug: 50 μg KIO-301 — KIO-301 drug product is an ophthalmic formulation of the drug substance KIO-300-Cl in sulfobutylether-β-cyclodextrin, sucrose, phosphate buffer salts and water suitable for IVT injection. The drug substance KIO-300-Cl is a quaternary ammonium chloride salt of the active compound KIO-300.
  Arms: 50 μg KIO-301

SUMMARY:
The goal of the study is to investigate the safety, tolerability and efficacy of up to 3 doses of KIO-301 administered by intravitreal (IVT) injection bilaterally every 6 weeks in patients with late-stage retinitis pigmentosa (RP).

Late-stage RP patients will include those patients with No Light Perception (NLP), or Low Vision (LV).

DETAILED DESCRIPTION:
All enrolled and randomised study participants will attend study visits every 3 weeks during treatment (12 weeks) and follow-up (12 weeks) for PK, safety, tolerability, and efficacy assessments. The Screening period may be up to 45 days. Total duration of the main study may be up to 30 weeks.

For participants who received placebo in the main study and choose to participate in the open label (OL) extension, duration of participation will be a further 24 weeks with total participation dependent upon time between completion of the main study and initiation of the OL extension.

ELIGIBILITY:
Inclusion Criteria:

1. Be aged 18 years or older at the time of consent.
2. Provide informed consent prior to any study procedures, as stipulated by local laws, Ethics Committee (EC) and Regulatory Authority (RA) guidelines.
3. Be willing and able to follow all study instructions, attend all study visits, and complete all study assessments.
4. Have a clinical diagnosis of non-syndromic RP, with the exception of Usher's Syndrome Type II (USH2) which is allowed.
5. Have a visual acuity as per the Berkeley Rudimentary Vision Test (BRVT) at Screening of:

   * NLP OU confirmed by inability to see pen torch light at 25 cm OD, OS, and OU (assigned logMAR of 4.0).
   * LV OU limited to logMAR > 1.6 and < 4.0.
6. Other than intravitreal corticosteroids, participants must not receive intravitreal concomitant medications from Screening until end of study.
7. For Low Vision (LV) OU participants only: must pass at least one multi-luminance functional vision (MLFV) test at two successive light levels (between 1 and 500 lux), or at 1400 lux. Additionally, they must fail the same test at 0.125 and 0.35 lux.
8. Must agree to follow appropriate contraception requirements from Screening until 3 months after the last dose of IMP.

   * Participants assigned female at birth who are of child-bearing potential (OCBP) must agree to a pregnancy test at Screening and use an acceptable method of birth control including oral, transdermal, injectable, or implantable hormonal contraception, intrauterine device, abstinence from intercourse with partner assigned male at birth, or surgical sterilisation of partner assigned male at birth. Participants assigned female at birth are not OCBP if they have had a hysterectomy, bilateral oophorectomy, bilateral tubal ligation, or are post-menopausal by at least 12 months.
   * Participants assigned male at birth with a partner OCBP must be surgically sterile for at least 3 months prior to starting study drug, or ensure their partner uses contraception as outlined above, and must use a male condom. Participants assigned male at birth must not donate sperm from Screening until 3 months after the last dose of IMP.
   * Participants who have practiced true abstinence for at least 1 year due to usual and preferred lifestyle choice are exempt from contraceptive requirements. If a participant who is abstinent becomes sexually active, they must agree to use appropriate contraception as described above.

Exclusion Criteria:

1. Pregnant or breast-feeding, or plan to become pregnant during the study.
2. Have, in the investigator's opinion, evidence of material/substantial optic nerve disease.
3. Have a history of one or more retinal detachments.
4. Other than RP related macular pathologies, have in the investigator's opinion, clinically significant ocular disease (e.g., corneal oedema, uveitis, severe keratoconjunctivitis sicca), or clinically significant opacities of the media which might interfere with the study assessments, or the ability of the participant to complete the study.
5. Have a history of high myopia (> 6 diopters).
6. Have uncontrolled severe glaucoma defined as intraocular pressure (IOP) of > 26 mmHg when on 2 or more IOP lowering medications and cup disc ratio of ≥ 0.8, as diagnosed by an ophthalmologist.
7. Have had a previous intraocular surgery (with the exception of phacoemulsification cataract surgery and YAG capsulotomy more than 12 months prior to first study drug administration, which is allowed).
8. Have aphakia or a subluxed intraocular lens, or have evidence of zonular weakness that in the opinion of the investigator would result in light obfuscation.
9. Have a psychiatric condition that, in the investigator's opinion, precludes compliance with the protocol; past or present psychoses; past or present bipolar disorder; disorder requiring lithium; or within five years prior to screening, a history of suicide plan.
10. Have any clinically significant abnormality at screening determined by medical history, vital signs, clinical biochemistry, haematology, urinalysis, or a 12-lead electrocardiogram (ECG), as assessed by the investigator, which might interfere with the study assessments or the ability of the participant to complete the study.
11. Have any other medical condition or significant co-morbidities, or any finding during screening, which in the view of the Investigator is likely to interfere with the study or put the Participant at risk, confound study data, or interfere significantly with study participation.
12. Have clinical signs of active ocular or systemic infection and/or a temperature greater than 38.0°C at the time of screening. Study entry must be deferred at least 14 days from resolution.
13. Have participated in any investigational study within 30 days prior to screening, prior exposure to an investigational product within 5 elimination half-lives, or planned used of an investigational product or device during the study.
14. Have known or suspected hypersensitivity to any of the study drug excipients.
15. Are taking any medications that are known to be toxic to the retina or optic nerve.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-08-29 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2027-08 (Estimated)

PRIMARY OUTCOMES:
To assess the safety and tolerability of multiple doses of KIO-301 administered by IVT injection bilaterally of KIO-301 in patients with late-stage RP. | Baseline (Week 1/pre-dose) to Week 25 (12 weeks post 3rd IVT administration of KIO-301)
  Change in ophthalmic and non-ophthalmic adverse events

CONTACTS AND LOCATIONS:
Overall Officials: Doron Hickey, MBChB, Principal Investigator — The Centre for Eye Research Australia (CERA); Robert Casson, MBBS (Hons), Principal Investigator — Royal Adelaide Hospital
Locations (5):
- Australia (5):
  - Save Sight Institute, Sydney, New South Wales
  - Queensland Eye Institute, Woolloongabba, Queensland
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Cerulea Clinical Trials, East Melbourne, Victoria
  - Lions Eye Institute, Nedlands, Western Australia

IPD SHARING:
Plan to Share IPD: Undecided